CLINICAL TRIAL: NCT00141466
Title: Cost Effectiveness of Two Different Implementation Procedures to Change Clinicians Practice Roles in the Detection of Hereditary Colorectal Cancer
Brief Title: Implementation of a New Strategy to Identify HNPCC Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: MIPA-2005; ZonMw nr. 945-14-107
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2008-04-23 (Estimated); Status verified 2007-02

CONDITIONS: Colorectal Neoplasms; Hereditary Nonpolyposis Colorectal Cancer
Keywords: Hereditary colorectal cancer; Microsatellite instability; Physician roles; Health care implementation; Intervention
MeSH Terms: conditions — Colorectal Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis; Microsatellite Instability | interventions — Educational Status

INTERVENTIONS:
Behavioral: Education for professionals
Behavioral: Distribution of educational materials
Behavioral: Feedback for professionals
Behavioral: Reminders for professionals

SUMMARY:
The purpose of this study is to compare two different strategies to implement a new method to identify patients with HNPCC, which appeared cost-effective and feasible. The effectiveness, costs and feasibility of both of the implementation strategies will be assessed.

DETAILED DESCRIPTION:
The Radboud University Nijmegen Medical Centre developed a new method to identify patients with HNPCC. This method appeared cost-effective and feasible. Using this new method 70% of the HNPCC patients will be identified as compared to less than 30% when the current method is used. However, this new method does not implement itself; large gaps exists between best evidence and daily practice. This study will compare an intensive strategy, consisting of distribution of educational materials, education, feedback and reminders, with a minimal strategy, only consisting of distribution of a critical care pathway. The aim is to find the most cost-effective strategy to implement the new method to identify patients with HNPCC in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer before the age of 50 years
* Second colorectal cancer at any age
* Colorectal cancer and other HNPCC associated extracolonic cancer irrespective of age at diagnosis
* Adenoma with high grade dysplasia diagnosed before the age of 40 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2005-09; Study Completion 2007-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of inclusion of eligible CRC-patients for MSI testing by pathologists.
Efficacy of referral of patients who are MSI positive to a clinical geneticist by surgeons.

SECONDARY OUTCOMES:
Experiences with and acceptance of changed physician practice roles by patients and clinicians.
Cost efficacy of the implementation procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Nicoline Hoogerbrugge, MD PhD, Principal Investigator — Department of Human Genetics, Radboud University Nijmegen Medical Center; Rosella P Hermens, MSc PhD, Principal Investigator — Center of Quality of Care Research, Radboud University Nijmegen Medical Center
Locations (13):
- Netherlands (13):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Meander Medisch Centrum, Amersfoort
  - Ziekenhuis Rijnstate, Arnhem
  - Pathologie laboratorium voor Dordrecht, Dordrecht
  - Stichting laboratoria voor pathologische anatomie en medische microbiologie, Eindhoven
  - Laboratorium voor pathologie Oost-Nederland, Enschede
  - Martini Ziekenhuis, Groningen
  - Elkerliek Ziekenhuis, Helmond
  - Laboratorium Volksgezondheid Friesland, Leeuwarden
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Medisch Centrum Rijnmond Zuid, Rotterdam
  - HagaZiekenhuis, The Hague
  - St. Elisabeth Ziekenhuis, Tilburg

REFERENCES:
- [Background] Kievit W, de Bruin JH, Adang EM, Severens JL, Kleibeuker JH, Sijmons RH, Ruers TJ, Nagengast FM, Vasen HF, van Krieken JH, Ligtenberg MJ, Hoogerbrugge N. Cost effectiveness of a new strategy to identify HNPCC patients. Gut. 2005 Jan;54(1):97-102. doi: 10.1136/gut.2004.039123. PMID 15591512
- [Background] de Bruin JH, Kievit W, Ligtenberg MJ, Nagengast FM, Adang EM, Ruers TJ, Kleibeuker JH, Sijmons RH, van Krieken JH, Hoogerbrugge N. [More hereditary intestinal cancer can be detected if patients with colorectal carcinoma that are selected by the pathologist are examined for microsatellite instability]. Ned Tijdschr Geneeskd. 2005 Aug 6;149(32):1792-8. Dutch. PMID 16121665
- [Derived] Overbeek LI, Hermens RP, van Krieken JH, Adang EM, Casparie M, Nagengast FM, Ligtenberg MJ, Hoogerbrugge N; MIPA study group. Electronic reminders for pathologists promote recognition of patients at risk for Lynch syndrome: cluster-randomised controlled trial. Virchows Arch. 2010 Jun;456(6):653-9. doi: 10.1007/s00428-010-0907-7. Epub 2010 Apr 9. PMID 20379742